CLINICAL TRIAL: NCT06518330
Title: Psychosis and Hallucinations in Methylphenidate-Treated Children: A Pharmacovigilance Study Using Vigibase
Brief Title: Psychosis Associated With Methylphenidate in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Caen_MPH_2024
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting a possible drug-induced adverse effects: Drug: search for methylphenidate intake
  Interventions: Drug: Intake of Methylphenidate

INTERVENTIONS:
Drug: Intake of Methylphenidate — Intake of Methylphenidate

SUMMARY:
perform a study in VigiBase® to assess if methylphenidate was associated with an over-reporting of psychosis including hallucinations in children and adolescents and to characterize those psychosis.

ELIGIBILITY:
Inclusion Criteria:

Case reported in the World Health Organization (WHO) database of individual safety case reports until 16/02/2024 in children and adolescents treated with drugs with an indication in ADHD.

Adverse events reported were including a list of MedDRA Preferred Terms related to psychosis

Exclusion Criteria:

Chronology not compatible between the drug and the toxicity

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with a possible drug-induced adverse effect
Sampling Method: Probability Sample
Enrollment: 46233 (Actual)
Dates: Start 1967-01-01 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Correlation between methylphenidate and psychosis in children and adolescents using a disproportionality analysis in Individual Case Reports involving at least one liable drug with an indication in ADHD. | from the 01/01/1967 to the 16/02/2024

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, France

IPD SHARING:
Plan to Share IPD: No